CLINICAL TRIAL: NCT06624436
Title: Immunomodulatory Effects of Dexamethasone, Tocilizumab and Anakinra During Experimental Human Endotoxemia
Acronym: DEDICATE-LPS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEDICATE-LPS; 2023-506556-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-20; First posted 2024-10-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-09

CONDITIONS: Sepsis; Neuroinflammatory Response; Immunosuppresion; Endotoxemia; Anakinra; Dexamethasone; Tocilizumab
Keywords: Sepsis; Immunosuppression; Systemic inflammation; Neuroinflammation; Anakinra; Dexamethasone; Tocilizumab; Human endotoxemia; Immunoparalysis; Hyperinflammatory response
MeSH Terms: conditions — Sepsis; Endotoxemia; Neuroinflammatory Diseases | interventions — Dexamethasone; tocilizumab; Interleukin 1 Receptor Antagonist Protein; Sodium Chloride; Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: DEDICATE-LPS is a randomized double-blind placebo-controlled (double-dummy) study. A total of 48 healthy male volunteers will undergo experimental human endotoxemia twice separated by one week. Volunteers will be randomized to an allocated study treatment (dexamethasone 6 mg i.v. (n = 12), tocilizumab 600 mg i.v. (n = 12), anakinra 200 mg i.v. (n = 12) or placebo (NaCl 0.9% i.v., n = 12)). Furthermore, 4 healthy male volunteers will be enrolled as a control group (receiving no study treatment or LPS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group 1: dexamethasone (Active Comparator): This arm (n = 12) of healthy male volunteers will have two LPS challenges (day 0 and day 7) and will receive dexamethasone infusion in 1 hour on the first LPS challenge.
  Interventions: Drug: Dexamethasone; Biological: LPS
- Group 2: Tocilizumab (Active Comparator): This arm (n = 12) of healthy male volunteers will have two LPS challenges (day 0 and day 7) and will receive Tocilizumab infusion in 1 hour on the first LPS challenge.
  Interventions: Drug: Tocilizumab; Biological: LPS
- Group 3: Anakinra (Active Comparator): This arm (n = 12) of healthy male volunteers will have two LPS challenges (day 0 and day 7) and will receive Anakinra infusion in 1 hour on the first LPS challenge.
  Interventions: Drug: Anakinra; Biological: LPS
- Group 4: Placebo (Placebo Comparator): This arm (n = 12) of healthy male volunteers will have two LPS challenges (day 0 and day 7) and will receive a placebo infusion in 1 hour on the first LPS challenge.
  Interventions: Drug: Placebo; Biological: LPS
- Group 5: Control (No Intervention): This arm (n = 4) of healthy male volunteers won't receive an LPS challenge or any of the study treatments. This group will be used to familiarise the study team with the study procedures and to establish the effect of placement of an intrathecal catheter on systemic and neuroinflammation.

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 6mg in 10mL NaCl 0.9% i.v. bolus + 100mL NaCl 0.9% placebo infusion in 1 hour on the first LPS challenge.
  Arms: Group 1: dexamethasone
Drug: Tocilizumab — Tocilizumab 600mg in 100mL NaCl 0.9% i.v. in 1 hour + a bolus of 10mL NaCl 0.9% placebo infusion on the first LPS challenge.
  Other Names: RoActemra; Tyenne
  Arms: Group 2: Tocilizumab
Drug: Anakinra — Anakinra 200mg in 100mL NaCl 0.9% i.v. in 1 hour + a bolus of 10mL NaCl 0.9% placebo infusion on the first LPS challenge.
  Other Names: Kineret
  Arms: Group 3: Anakinra
Drug: Placebo — Bolus of 10mL NaCl 0.9% placebo + 100mL NaCl 0.9% placebo infusion in 1 hour on the first LPS challenge.
  Other Names: NaCl 0.9%
  Arms: Group 4: Placebo
Biological: LPS — This is a non-investigational product. It is used as challenge agent to achieve a controlled inflammatory state.
  Other Names: Endotoxin; Lipopolysaccharide (LPS from E. coli type O113)
  Arms: Group 1: dexamethasone; Group 2: Tocilizumab; Group 3: Anakinra; Group 4: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the immunomodulatory effects of the drugs dexamethasone, tocilizumab and anakinra in healthy male subjects aged 18 to 35 undergoing experimental endotoxemia. The main questions it aims to answer are:

* What are the effects of these drugs on the development of immunoparalysis in a repeated human endotoxemia model?
* What is the extent of the neuroinflammatory response and how do these drugs affect neuroinflammation in a repeated human endotoxemia model?

Researchers will compare these drugs to a placebo (a look-alike substance that contains no drug).

Participants will visit the Intensive Care research department on two or five occasions (screening included):

* The intervention group will receive an LPS challenge twice, with a week in between. Before the first LPS challenge, one of the described drugs will be administered. Blood, saliva and tear fluid will be collected regularly during the LPS challenge. Cerebrospinal fluid will also be collected through a catheter in the spinal cord.
* The control group will not receive an LPS challenge or drug administration and will have only one study day. During this day, blood, saliva, tear fluid and cerebrospinal fluid will be collected as regularly as during the LPS challenge of the intervention group.

During an LPS challenge, the investigators mimic blood poisoning by giving an endotoxin, also called LPS. This is a small part of the cell wall of a bacteria. This will cause transient flu-like symptoms for 3-4 hours.

DETAILED DESCRIPTION:
The experimental human endotoxemia model is a controlled, standardized and safe model of systemic (sepsis-like) inflammation induced by bacterial lipopolysaccharide (LPS) in healthy volunteers. This model captures many hallmarks of both the hyperinflammatory phenotype (observed following a first LPS challenge) and the immunoparalytic phenotype (observed following a second LPS challenge one week later) of sepsis.

In this study the investigators aim to determine the effects of dexamethasone, tocilizumab and anakinra within the repeated experimental human endotoxemia model on the development of immunoparalysis, reflected by between-group differences in plasma TNF (and other cytokine) concentrations upon the second LPS challenge. The investigators will also profile inflammatory parameters in cerebrospinal fluid (CSF), reflected by within- and between-group differences in CSF TNF (and other cytokine) concentrations following the first LPS challenge, to gain insights in inflammatory responses of the central nervous system.

Anti-inflammatory drugs may help reduce sepsis-induced immunoparalysis and, somewhat counterintuitively, improve immune responses later by dampening the initial hyperinflammation. Pro-inflammatory cytokines, such as TNF, are key in triggering this immunosuppression. Reducing early hyperinflammation could also prevent postoperative immune suppression, lowering the risk of infections. Drugs like dexamethasone, tocilizumab, and anakinra may affect neuroinflammation, depending on their ability to cross the blood-brain barrier (BBB).

Furthermore, the investigators will explore whether cytokine profiles in saliva and tear fluid can be used as a proxy for circulating cytokine responses. Saliva and tear fluid cytokines may serve as non-invasive alternatives to blood measurements, especially for vulnerable populations, though more research is needed to validate their reliability.

Comprehensive assessment of cellular components and cytokine dynamics in blood, CSF, saliva, and tear fluid will be conducted using RNA sequencing, providing insights into cellular and molecular mechanisms during endotoxemia and drug effects. This research will help identify new drug targets and better understand the immunomodulatory effects of dexamethasone, tocilizumab, and anakinra on inflammation and immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥18 and ≤35 years
* Body mass index (BMI) ≥18 and ≤30 kg/m2
* Healthy (as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram and routine clinical laboratory parameters)
* Able to comprehend and sign the Information letter and Informed Consent (IC) prior to enrolment in the study.

Exclusion Criteria:

* Use of any prescription medication or over-the-counter non-steroidal anti-inflammatory drugs
* Known anaphylaxis or hypersensitivity to any (non-)investigational products or their excipients
* History of chronic headache or previous post-dural puncture headache (PDPH)
* History or signs of severe atopic syndrome (asthma, rhinitis with medication and/or eczema)
* History of any disease associated with immune deficiency
* History of cancer in the last 5 years (excluding localised skin cancer or carcinoma in situ)
* History or signs of haematological disease
* History or signs of thromboembolic disorders
* History of peptic / gastric ulcer disease
* History of psychiatric disorders
* Thrombocytopenia (<150*109/mL) or anaemia (<8.0 mmol/L)
* History, signs or symptoms of cardiovascular disease, in particular:

  * Prone to vagal collapse
  * History of atrial or ventricular arrhythmia
  * Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrio-ventricular block or a complete left bundle branch block
  * Hypertension (defined as RR systolic > 160 or RR diastolic > 90 mmHg)
  * Hypotension (defined as RR systolic < 100 or RR diastolic < 50 mmHg)
* Renal impairment (defined as plasma creatinine >120 μmol/L)
* Liver enzyme abnormalities (above 2x the upper limit of normal)
* Signs of infection (CRP > 20 mg/L, white blood cells > 12x109/L or

  * lt; 4x109/L)
* Clinically significant acute illness, including infections or trauma, within 1 month prior to the first LPS challenge
* Previous (participation in a study with) endotoxin (LPS) administration
* Participation in an experimental intervention or drug trial within 3 months prior to the first LPS challenge
* Any vaccination or blood donation within 1 month prior to the first LPS challenge
* Recent hospital admission or surgery with general anaesthesia within 3 months prior to the first LPS challenge
* Use of recreational drugs within 2 weeks prior to the first LPS challenge
* Suspected of not being able to comply with the trial protocol
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Between-group differences in plasma TNF concentrations upon the second LPS challenge | 1 day (during second LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the development of immunoparalysis in a repeated endotoxemia model in humans, reflected by between-group differences in plasma TNF concentrations upon the second LPS challenge.
Within and between-group differences in CSF TNF concentrations during repeated experimental human endotoxemia | 8 days
  The extent of the neuroinflammatory response as well as the effects of dexamethasone, tocilizumab and anakinra on neuroinflammation, reflected by within and between-group differences in CSF TNF concentrations during repeated experimental human endotoxemia

SECONDARY OUTCOMES:
Between-group differences in plasma cytokine concentrations during the second LPS challenge (e.g. IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10, CX3CL1, YKL-40). | 1 day (during the second LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the development of systemic immunoparalysis as reflected by plasma concentrations of other mediators than TNF (e.g. IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10, CX3CL1, YKL-40) during the second LPS challenge.
Between-group differences in the log2-fold change of the Area Under the Curves (AUCs) of plasma cytokine concentrations (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10, CX3CL1, YKL-40) during the first and second LPS challenges. | 8 days
  The effects of dexamethasone, tocilizumab and anakinra on the development of systemic immunoparalysis as reflected by between-group differences in the log2-fold change of the Area Under the Curves (AUCs) of plasma concentrations of other mediators than TNF during the first and second LPS challenges.
Between-group differences in other plasma inflammatory proteins upon the second LPS challenge, as measured by the Olink Target 96 inflammation panel (92 protein biomarkers). | 1 day (during the second LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the development of systemic immunoparalysis as measured by the Olink Target 96 inflammation panel (92 protein biomarkers) upon the second LPS challenge.
Between-group differences in the log2-fold change of peak plasma concentrations of other inflammatory proteins, as measured by the Olink Target 96 inflammation panel (92 protein biomarkers), during the first and second LPS challenges | 8 days
  The effects of dexamethasone, tocilizumab and anakinra on the development of systemic immunoparalysis as measured by the Olink Target 96 inflammation panel (92 protein biomarkers), during the first and second LPS challenges.
Between-group differences in mHLA-DR during the first and second LPS challenge. | 8 days
  The effects of dexamethasone, tocilizumab and anakinra on the development of systemic immunoparalysis as reflected by between-group differences in mHLA-DR during the first and second LPS challenge.
Between-group differences in plasma cytokine concentrations during the first LPS challenge (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10, CX3CL1, YKL-40). | 1 day (during the first LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the acute systemic inflammatory response during the first LPS challenge as reflected by between-group differences in plasma cytokine concentrations (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10, CX3CL1, YKL-40).
Between-group differences in other plasma inflammatory proteins upon the first LPS challenge, as measured by the Olink Target 96 inflammation panel (92 protein biomarkers). | 1 day (during the first LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the acute systemic inflammatory response during the first LPS challenge as measured by the Olink Target 96 inflammation panel (92 protein biomarkers).
Between-group differences in symptom scores during the first LPS challenge. | 1 day (during the first LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the acute systemic inflammatory response during the first LPS challenge as reflected by between-group differences in symptom scores.
Between-group differences in blood pressure during the first LPS challenge. | 1 day (during the first LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the acute systemic inflammatory response during the first LPS challenge as reflected by between-group differences in blood pressure.
Between-group differences in temperature during the first LPS challenge. | 1 day (during the first LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the acute systemic inflammatory response during the first LPS challenge as reflected by between-group differences in temperature.
Between-group differences in heart rate during the first LPS challenge. | 1 day (during the first LPS challenge)
  The effects of dexamethasone, tocilizumab and anakinra on the acute systemic inflammatory response during the first LPS challenge as reflected by between-group differences in heart rate.
Within and between-group differences in blood leukocyte single cell and/or bulk mRNA profiles/transcriptomic pathways upon both LPS challenges. | 8 days
  The effects of LPS-induced inflammation, dexamethasone, tocilizumab and anakinra on transcriptome profiles of circulating leukocytes during the first and second LPS challenges.
Within and between-group differences in cytokine production of leukocyte cultures | 8 days
  The effects of dexamethasone, tocilizumab and anakinra on ex vivo leukocytic cytokine production
Within and between-group differences in plasmatic coagulation parameters (e.g. whole blood thrombin generation and plasma thrombin generation) upon both LPS challenges. | 8 days
  The effects of dexamethasone, tocilizumab and anakinra on plasmatic coagulation, as reflected by within and between-group differences in thrombin generation during the first and second LPS challenges.
Within and between-group differences in CSF cytokine concentrations during both LPS challenges (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G CSF, IP-10, CX3CL1, YKL-40, HSP-70, Aß-40, Aß-42, pTau, NfL). | 8 days
  The effects of LPS administration as well as dexamethasone, tocilizumab and anakinra on neuroinflammation during the first and second LPS challenges as reflected by within and between-group differences in CSF cytokine concentrations (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G CSF, IP-10, CX3CL1, YKL-40, HSP-70, Aß-40, Aß-42, pTau, NfL).
Within and between-group differences in other inflammatory proteins in CSF upon both LPS challenges, measured by the Olink Target 96 inflammation panel (92 protein biomarkers). | 8 days
  The effects of LPS administration as well as dexamethasone, tocilizumab and anakinra on neuroinflammation during the first and second LPS challenges, as reflected by within and between-group differences in other inflammatory proteins in CSF, measured by the Olink Target 96 inflammation panel (92 protein biomarkers).
Between-group differences in the log2-fold change of the AUCs of CSF cytokine concentrations during the first and second LPS challenges. | 8 days
  The effects of LPS administration as well as dexamethasone, tocilizumab and anakinra on neuroinflammation during the first and second LPS challenges as reflected by within and between-group differences in the log2-fold change of the AUCs of CSF cytokine concentrations during the first and second LPS challenges.
Within and between-group differences in CSF leukocyte single cell and/or bulk mRNA profiles/transcriptomic pathways upon both LPS challenges. | 8 days
  The effects of LPS-induced inflammation, dexamethasone, tocilizumab and anakinra on transcriptome profiles of cells in the CSF during the first en second LPS challenges.
Correlation between systemic and CSF markers during systemic inflammation upon both LPS challenges (e.g. cytokines, Olink, transcriptome profiles). | 8 days
  The relationship between systemic inflammatory responses and neuroinflammation as reflected by the correlation between systemic and CSF markers during systemic inflammation during the first en second LPS challenges (e.g. cytokines, Olink, transcriptome profiles).
Concentrations of dexamethasone, anakinra and tocilizumab in blood and CSF upon both LPS challenges. | 8 days
  The pharmacokinetics of dexamethasone, tocilizumab and anakinra in blood and CSF during LPS-induced inflammation.
Kel (elimination rate constant) of dexamethasone, anakinra and tocilizumab in blood and CSF upon both LPS challenges. | 8 days
  The pharmacokinetics of dexamethasone, tocilizumab and anakinra in blood and CSF during LPS-induced inflammation.
Tmax (time at maximum concentration) of dexamethasone, tocilizumab and anakinra in blood and CSF upon both LPS-challenges. | 8 days
  The pharmacokinetics of dexamethasone, tocilizumab and anakinra in blood and CSF during LPS-induced inflammation.
Cmax (maximum concentration) of dexamethasone, anakinra and tocilizumab in blood and CSF upon both LPS challenges. | 8 days
  The pharmacokinetics of dexamethasone, tocilizumab and anakinra in blood and CSF during LPS-induced inflammation.
AUCs (area under the curves) of dexamethasone, anakinra and tocilizumab in blood and CSF upon both LPS challenges. | 8 days
  The pharmacokinetics of dexamethasone, tocilizumab and anakinra in blood and CSF during LPS-induced inflammation.
T1/2 (terminal elimination half-life) of dexamethasone, anakinra and tocilizumab in blood and CSF upon both LPS challenges. | 8 days
  The pharmacokinetics of dexamethasone, tocilizumab and anakinra in blood and CSF during LPS-induced inflammation.

OTHER OUTCOMES:
Within and between-group differences in cytokine concentrations in saliva and tear fluid during both LPS challenges (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10). | 8 days
  The effects of LPS administration as well as dexamethasone, tocilizumab and anakinra on salivary and tear fluid cytokine levels, as reflected by within and between-group differences in cytokine concentrations (e.g. TNF, IL1RA, IL-6, IL-8, IL-10, MIP-1α, MIP-1ß, MCP-1, G-CSF, IP-10) during the first and second LPS challenges.
Correlation between cytokines in plasma, saliva, and tear fluid during systemic inflammation upon both LPS challenges. | 8 days
  The relationship between systemic, salivary and tear fluid cytokine responses as reflected by the correlation between cytokines in plasma, saliva, and tear fluid during systemic inflammation during the first and second LPS challenges.
Within and between-group differences in single cell and/or bulk mRNA profiles/transcriptomic pathways of cells in saliva upon both LPS challenges. | 8 days
  The effects of LPS-induced inflammation, dexamethasone, tocilizumab and anakinra on transcriptome profiles of cells in saliva, as reflected by within and between-group differences in single cell and/or bulk mRNA profiles/transcriptomic pathways of cells during the first and the second LPS challenges.
Within and between-group differences in single cell and/or bulk mRNA profiles/transcriptomic pathways of cells in tear fluid upon both LPS challenges. | 8 days
  The effects of LPS-induced inflammation, dexamethasone, tocilizumab and anakinra on transcriptome profiles of cells in tear fluid, as reflected by within and between-group differences in single cell and/or bulk mRNA profiles/transcriptomic pathways of cells during the first and the second LPS challenges.
Number of adverse events related to the use of dexamethasone, tocilizumab and anakinra. | 8 days
  Safety of dexamethasone, tocilizumab and anakinra as reflected by the number of adverse events related to their use.
Correlation of blood nitric oxide concentrations between exercise, stress and inflammation. | Upon the screening day and both LPS challenges (3 days)
  The kinetics of blood nitric oxide concentrations during exercise (bicycling on a home-trainer during screening), stress and systemic inflammation (during the first and second LPS challenges).

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
* Demographic data (pseudonimized)
  * Outcome data (pseudonimized)
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning directly after publication of the paper describing the main results of the study and ending 30 years after publication of the paper describing the main results.
Access Criteria: Data will be made available upon reasonable request to the corresponding author.